CLINICAL TRIAL: NCT03128515
Title: Optimizing Hydroxyurea Therapy in Children With Sickle Cell Anemia In Malaria Endemic Areas: The NOHARM Maximum Tolerated Dose (MTD) Study
Brief Title: Optimizing Hydroxyurea Therapy in Children With SCA In Malaria Endemic Areas
Acronym: NOHARM-MTD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Makerere University (Other); Mulago Hospital, Uganda (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Chandy John, Professor of Pediatrics, Medicine, Microbiology and Immunology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00456728
Record Dates: First submitted 2017-03-22; First posted 2017-04-25 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease; Malaria
Keywords: Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell; Malaria | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTD Dose Escalation (Experimental): Maximum tolerated dose of Hydroxyurea, 25-30 mg/kg/day
  Interventions: Drug: Hydroxyurea
- Fixed Dose (Active Comparator): Fixed dose of Hydroxyurea, 20 mg/kg/day
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Administered once a day in tablet form (100mg or scored 1000mg) for 24 months
  Other Names: Siklos; Hydroxycarbamide

SUMMARY:
The Novel use Of Hydroxyurea in an African Region with Malaria (NOHARM) study is the first placebo-controlled randomized clinical trial of hydroxyurea treatment in a malaria endemic region. NOHARM has now achieved full enrollment; all children have completed the blinded portion of the protocol and are in the open-label study treatment portion.

This extension study of maximum tolerated dose (MTD), addresses the next critical set of questions about the optimal dosing and monitoring of hydroxyurea treatment for children with SCA in low-resource settings. By providing guidance about optimal hydroxyurea treatment, the NOHARM MTD Study will directly inform policies that can transform the health of African children living with SCA.

DETAILED DESCRIPTION:
All children enrolled in NOHARM received hydroxyurea treatment at a fixed daily dose of 20 mg/kg/day. This dose was selected as a likely safe dose, but does not escalate hydroxyurea to MTD as is commonly done in the US. Without this information, we cannot know whether hydroxyurea treatment at the MTD would be feasible (since it requires closer monitoring to avoid hematological toxicities), safe (since adverse events may be greater with MTD, risk of malaria may be altered by MTD, and risk of infections as a result of neutropenia could also be greater with MTD) or beneficial (MTD is associated with higher hemoglobin and fetal hemoglobin concentration).

In this extension MTD study of open-label hydroxyurea for children in NOHARM who complete the initial study, consented children will be randomized to either fixed-dose or MTD hydroxyurea treatment for a minimum of 24 months. If hydroxyurea treatment continues to prove safe and effective in this low-resource malaria endemic area, and an optimal dosing scheme is determined, then the long-term goal is for all study children to transition to hydroxyurea treatment provided through the Ugandan Ministry of Health. To provide for a smooth transition, we will continue all children at either MTD or fixed dose hydroxyurea until a common end date (November 2019), at which time all study participants will have received a minimum of 24 months of additional hydroxyurea (either MTD or fixed dose). Addmedica, the Paris-based pharmaceutical company that provides the current active drug and placebo for the NOHARM trial, has agreed to provide additional hydroxyurea for this MTD study at no cost to the study or the participants.

The Specific Aims of the NOHARM MTD proposal include two initiatives for participants who are currently enrolled in NOHARM:

Aim 1. To determine the safety and efficacy of maximum tolerated dose (MTD) vs. fixed dose (20 mg/kg/day) hydroxyurea treatment in children with SCA in a low-resource, malaria endemic setting. For safety, we will compare adverse events and severe adverse events, including hematologic toxicities. For efficacy, we will assess hemoglobin level, fetal hemoglobin percentage (% HbF), and incidence of vaso-occlusive events such as pain crisis and acute chest syndrome.

Aim 2. To compare the clinical outcomes of MTD vs. fixed dose hydroxyurea treatment in children with SCA in a low-resource, malaria endemic setting. Clinical outcomes assessed will include growth and malaria incidence over a 24-month follow-up period, and differences in renal, splenic, and cerebrovascular function between study entry and 24-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children with confirmed SCA who participated in the NOHARM study of hydroxyurea at the Mulago Hospital Sickle Cell Clinic (MHSCC), will be eligible for the MTD study after completing both 12-months of blinded study treatment and then an additional 12-months of open-label hydroxyurea for the second year of the study.
* The age range for enrollment into NOHARM, which began in 2014, was 1-4 years. Therefore, the children who will be enrolled in the follow up MTD study will be 3-6 years of age.

Exclusion Criteria:

* Not willing to come for all scheduled clinical visits or accept randomization

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2019-04-07 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Proportion of children with average hemoglobin ≥9.0 g/dL or average HbF ≥20% | Over 24 month period on study drug
  Proportion of children who achieve either an average hemoglobin ≥9.0 g/dL or an average HbF ≥20% after 24 months on study drug

SECONDARY OUTCOMES:
Clinical malaria incidence | Over 24 month period on study drug
  Clinical malaria is defined as a history of fever or measured axillary temperature ≥37.5 degrees, plus Plasmodium species on blood smear.
Vaso-occlusive crises | Over 24 month period on study drug
  SCA-related adverse events defined as:
  * Pain event
  * Dactylitis
  * Acute chest syndrome
Incidence of severe adverse events (SAE) | Over 24 month period on study drug
  Death, hospitalization >7 days, life-threatening event
Incidence of hematologic toxicities | Over 24 month period on study drug
  Hematologic toxicities are defined as:
  * Hemoglobin (Hb) <4.0g/dL
  * Hb <6.0g/dL AND absolute reticulocyte count (ARC) <100 x 10E9/L
  * Hb <7.0g/dL AND ARC <80 x 10E9/L
  * Platelets <80 x 10E9/L
  * Absolute neutrophil count (ANC) <1.0 x 10E9/L
Cerebrovascular function | At study treatment initiation then at 12 months and 24 months after study initiation
  Transcranial Doppler blood vessel velocity to determine cerebrovascular function
Change in creatinine levels | Over 24 month period on study drug
  Changes in creatinine level as a measure of renal function
Change in cystatin C | Over 24 month period on study drug
  Changes in cystatin C level as a measure of renal function
Change in splenic function | Over 24 month period on study drug
  Quantitative micronuclei [Howell Jolly bodies] measured by flow cytometry
Change in height-for-age z-score | Over 24 month period on study drug
  Change in height-for-age z-score
Change in weight-for-age z-score | Over 24 month period on study drug
  Change in weight-for-age z-score
Change in weight-for-height z-score | Over 24 month period on study drug
  Change in weight-for-height z-score

CONTACTS AND LOCATIONS:
Overall Officials: Chandy C John, M.D., Principal Investigator — Indiana University
Locations (1):
- Mulago Hospital Sickle Cell Clinic, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] John CC, Opoka RO, Latham TS, Hume HA, Nabaggala C, Kasirye P, Ndugwa CM, Lane A, Ware RE. Hydroxyurea Dose Escalation for Sickle Cell Anemia in Sub-Saharan Africa. N Engl J Med. 2020 Jun 25;382(26):2524-2533. doi: 10.1056/NEJMoa2000146. PMID 32579813